CLINICAL TRIAL: NCT06385054
Title: Effect of Probiotics on Infantile Colic Symptoms: a Randomized, Double-blind, Placebo-controlled Study (EPIC).
Brief Title: Effect of Probiotics on Infantile Colic Symptoms
Acronym: EPIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lallemand Health Solutions (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: L-027; 2023-A02612-43 (Registry Identifier: ID-RCB); PEC23063 (Other: Biofortis)
Record Dates: First submitted 2024-04-23; First posted 2024-04-25 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Infantile Colic
Keywords: EPIC; Infant Colic; Probiotics; Crying Time; Gut Microbiota; Sleep Duration
MeSH Terms: conditions — Colic | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Participants in this group will be randomized to receive the probiotic B. lactis B94 for 4 weeks.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Participants in this group will be randomized to receive a placebo for 4 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Participants will be taking 1 sachet a day, at a similar time every day, dissolved in 10 ml of lukewarm water.
  Arms: Probiotic
Dietary Supplement: Placebo — Participants will be taking 1 sachet a day, at a similar time every day, dissolved in 10 ml of lukewarm water.
  Arms: Placebo

SUMMARY:
The aim of this clinical trial is to assess the impact of B. lactis B94 on participants with infantile colic. It is hypothesized that participants given the probiotic formula will have a significant reduction in their crying duration compared to participants receiving the placebo, after 4 weeks of intervention.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the potential beneficial effects of B. lactis B94 on the symptoms of infantile colic.

Participants diagnosed with infantile colic will be recruited to participate in this randomized, double-blind, placebo controlled, two-armed parallel study. Eligible participants will be enrolled in this study for 6 weeks, and will undergo a 1-week run-in baseline period followed by a 4-week interventional period, then a 1-week follow-up period.

The study will consist of 3 in-person visits and 4 phone calls.

ELIGIBILITY:
Inclusion Criteria:

I1. Healthy male or female. I2. Age ≤ 8 weeks old. I3. Diagnosis of infantile colic according to the Rome IV criteria. Infants must show cry or fuss behavior for 3 or more hours per day, during 3 or more days in 7 days.

I4. Exclusively breastfeeding and planning to breastfeed for the duration of the study.

I5. With a written informed consent signed by the father and mother or legal guardian.

I6. With parents willing to complete questionnaires, records, and diaries associated to the study and to complete all clinical visits and scheduled telephone calls.

I7. At least one of the legal representatives is affiliated with a social security scheme.

Exclusion Criteria:

E1. Birthweight < 2500 g. E2. Gestational age < 37 weeks. E3. Apgar score at 5 minutes < 7. E4. Partially or fully formula fed infants except for the 4 first days after birth.

E5. Stunted growth/weight loss (< 100 g/week from birth to last reported). E6. Gastroesophageal reflux disease, short bowel syndrome, chronic intestinal diseases, or gastrointestinal malformations.

E7. Diagnosed or reported fever and/or infectious diseases, or current systemic infections, or history of congenital infections.

E8. Genetic diseases and chromosomal abnormalities. E9. Metabolic diseases or pancreatic insufficiency. E10. Immunodeficiency. E11. Neurological diseases. E12. Suspected or confirmed food allergies and intolerances. E13. Mother who consumed antacid medications (proton pump inhibitor and H2 receptor antagonist) within the month before birth and intend to consume any during the trial.

E14. Use of probiotics, prebiotics, antibiotics, or gastric acid inhibitors by the infant at any time from birth to the moment of screening and during the trial.

E15. Use of anti-colic medication at any time from birth to the moment of screening.

E16. Use of probiotics and prebiotics supplements by the mother between the birth of their infant and the moment of screening and intend to consume any during the trial.

E17. Currently enrolled in another clinical study or having participated in another clinical from birth to the moment of screening.

E18. Whose legal representatives have psychological or linguistic incapability to sign the informed consent.

E19. Impossibility to contact the legal representatives in case of emergency.

Max Age: 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in daily crying duration | 4 weeks
  Proportion of infants who experience a decrease of mean daily crying duration of at least 50% after 4 weeks of intervention, in placebo versus probiotic groups.

SECONDARY OUTCOMES:
Change in crying patterns | 4 weeks
  Proportion of infants who experience a decrease of mean daily crying duration of at least 50% or at least 25%, mean daily number of crying episodes and variation in mean daily crying duration after 1, 2, 3, 4 weeks of intervention, in placebo versus probiotic groups.
Change in sleep duration | 4 weeks
  Variation in the mean daily duration of the infant's sleep after 1, 2, 3, 4 weeks of intervention in probiotic versus placebo groups.
Change in maternal quality of life | 4 weeks
  Variation in the maternal score of the mother quality-of-life questionnaire (SF- 36) after 4 weeks of intervention in probiotic versus placebo groups.
Change in bowel habits | 4 weeks
  General perception of colic evolution (total recovery / better / worse / no change), infant bowel movement frequency (mean daily number of stools) and stool consistency (rate (%), Amsterdam infant stool scale) after 1, 2, 3, 4 weeks of intervention in probiotic versus placebo groups.
Change in gut microbiota composition | 4 weeks
  Gut microbiota composition (α-diversity, β-diversity, and relative abundance at the genus level) and variation in gut microbiota composition (α-diversity, β-diversity, and relative abundance at the genus level) after 4 weeks of intervention in probiotic versus placebo groups (via 16S sequencing).
Probiotic strain recovery | 4 weeks
  Recovery of the probiotic strain in infant stool samples (qPCR) after 4 weeks of intervention.

OTHER OUTCOMES:
Safety and tolerability of the intervention | 5 weeks
  Assessment of the safety and tolerability of the probiotic formulation and the placebo through records of AEs/SAEs, growth parameters and number of unscheduled visits to the doctor.
Change in fecal immune markers and proteins | 4 weeks
  Difference in the concentration of fecal immune markers and proteins after 4 weeks of intervention in probiotic versus placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Pr. Nicholas Kalach, MD, Principal Investigator — Groupement des Hôpitaux de l'Institut Catholique de Lille
Locations (10):
- France (10):
  - Cabinet privé Dr Regimbart-Trubuil Christine, Bécon-les-Granits
  - Centre Hospitalier de Boulogne-sur-Mer, Boulogne-sur-Mer
  - CHU Caen Normandie, Caen
  - CHU Grenoble Alpes, La Tronche
  - Hôpital Saint Vincent de Paul, Lille
  - Centre Hospitalier de Montauban, Montauban
  - CHU de NANTES, Nantes
  - Biofortis, Unité d'investigation Clinique, Paris
  - Biofortis, Unité d'investigation Clinique, Saint-Herblain
  - Centre Hospitalier du val d'Ariège, Saint-Jean-de-Verges

IPD SHARING:
Plan to Share IPD: No